CLINICAL TRIAL: NCT01730001
Title: A Prospective Randomized Controlled Trial Comparing Competent EARLY-intubation to LATE-intubation in Patients With Prehospital GCS < 9 and Short Transport Time to Hospital.
Brief Title: Early Versus Late Intubation Trial in Physician Manned Emergency Medical Services
Acronym: ELITE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn, no patients included
Sponsor: Norwegian Air Ambulance Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLA-3104-03/04
Record Dates: First submitted 2012-11-10; First posted 2012-11-21 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Trauma; Craniocerebral Trauma; Intracerebral Hemorrhage; Seizures; Unconsciousness
MeSH Terms: conditions — Wounds and Injuries; Craniocerebral Trauma; Cerebral Hemorrhage; Seizures; Unconsciousness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Intubation (Active Comparator): Early intubation is defined as prehospital intubation on the scene of the patient illness/injury, or where the EMS physician first meets the patient (e.g en route to hospital). Intubation includes drug assisted and/or rapid sequence intubation (RSI) with endotracheal tube.
  Interventions: Procedure: Early Intubation
- Late intubation (Active Comparator): Late intubation is defined as on-scene prehospital high-flow (> 10 L/min) supplemental oxygen by mask, assisted bag-mask-ventilation by EMS physician if required and stable recovery position during transport to hospital. Intubation should be done on arrival in the emergency department.
  Interventions: Procedure: Late intubation

INTERVENTIONS:
Procedure: Early Intubation
  Arms: Early Intubation
Procedure: Late intubation
  Arms: Late intubation

SUMMARY:
This study looks at advanced airway management in critically ill or injured patients treated by physician manned emergency medical services, comparing early (on-scene) intubation to late (emergency department) intubation.

DETAILED DESCRIPTION:
The ELITE trial is a prospective randomized controlled trial (RCT) to compare competent EARLY-intubation to LATE-intubation in patients with on-scene Glasgow Coma Scale (GCS) < 9 and short ambulance transport times (< 20 min) to hospital.

The study aims to establish if advanced airway management with endotracheal intubation (ETI) in the field by specially trained Emergency Medical Services (EMS) physicians - compared to endotracheal intubation (ETI) performed by physicians in the emergency department in the same group - improves outcome in terms of 30-day mortality, degree of disability at discharge, complications and length of hospital stay, and neurologic outcome at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years)
* Initial GCS < 9 independent of cause.
* Intact airway reflexes and no impending airway obstruction.
* Located < 20 min ambulance transport time from nearest hospital emergency department.

Exclusion Criteria:

* Pediatric patients (under 18 years).
* Primary cardiorespiratory arrest (of non-traumatic / medical cause).
* Planned helicopter transport to hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01-01 (Estimated); Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
30 days mortality after injury or illness. | 30 days after illness or injury
  Dead or alive
Neurologic outcome at 6 months after injury or illness. | 6 months after illness or injury
  Neurologic outcome will be assessed using glascow outcome scores (GOS-E)

SECONDARY OUTCOMES:
Intubation success rates and airway management complications for the entire cohort and for key subsets | up to 6 months after illness or injury
Length of hospital stay, complications and degree of disability at discharge. | up to 6 months after illness or injury
Prevalence of adverse effects like cardiovascular complications (e.g. bradycardia, hypotension, asystole), and respiratory complications (e.g. hypoxia, pneumothorax). | up to 6 months after illness or injury

CONTACTS AND LOCATIONS:
Overall Officials: Geir A Sunde, MD, Principal Investigator — Norwegian Air Ambulance Foundation; Stephen JM Sollid, MD, PhD, Ass.Prof, Study Chair — Norwegian Air Ambulance Foundation; Hans M Lossius, MD, PhD, Prof, Study Director — Norwegian Air Ambulance Foundation; Espen Fevang, MD, Principal Investigator — Norwegian Air Ambulance Foundation
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Norwegian Air Ambulance Foundation, Drøbak

REFERENCES:
- See also: Norwegian Air Ambulance Foundation — http://www.norskluftambulanse.no